CLINICAL TRIAL: NCT00803088
Title: A Multicenter Clinical Trial Evaluating the Safety of Bronchial Thermoplasty Performed With the Alair® System During Two Treatment Sessions to Treat Severe Asthma.
Brief Title: Safety of Bronchial Thermoplasty Performed With the Alair® System During Two Treatment Sessions to Treat Severe Asthma
Acronym: 3to2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Current treatment regimen of 3 procedures considered acceptable.
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-01
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Treatment of airways with the Alair System
  Interventions: Device: The Alair System

INTERVENTIONS:
Device: The Alair System — Treatment of airways with the Alair System

SUMMARY:
The objective of this multicenter, single-arm, open-label clinical study is to evaluate the safety of performing bronchial thermoplasty with the Alair® System during two treatment sessions to treat severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult between the ages of 18 to 70 years.
* Subject is able to read, understand, and sign a written Informed Consent form to participate in the Study.
* Subject has asthma and is taking maintenance asthma medication that includes:

  1. Inhaled corticosteroid (ICS) at a dosage ≥1000μg beclomethasone per day or equivalent, AND long acting β2-agonist (LABA) at a dosage of ≥100μg per day Salmeterol or equivalent.
  2. Other asthma medications such as leukotriene modifiers, or anti-IgE, are acceptable (Subjects on Xolair® must have been on Xolair for greater than 1 year).
  3. Oral corticosteroids (OCS) at a dosage up to, but not greater than, 10mg per day.
* Subject has an AQLQ score at Baseline of 6.25 or less.
* Subject has a Pre-bronchodilator FEV1 of greater than or equal to 60% of predicted after medication stabilization during the Baseline Period.
* Subject has a PC20 < 8mg/ml per methacholine inhalation test using standardized methods*.
* Subject has at least one day of asthma symptoms during the 2 weeks of the Baseline Diary Period.
* Subject is a non-smoker for 1 year or greater (if former smoker, less than 10 pack years total smoking history).
* Subject is able to undergo bronchoscopy in the opinion of the Investigator or per hospital guidelines.
* Subject is willing and able to comply with the Study protocol, attending follow-up visits, and requirements for taking and abstaining from medications.

Exclusion Criteria:

* Subject participated in another clinical trial within 6 weeks of the Baseline Period involving respiratory intervention that could affect the outcome measures of this Study.
* Subject requirement during the Baseline Diary period for rescue medication use other than for prophylactic use for exercise exceeds an average of:

  1. 8 puffs per day of short-acting bronchodilator, or
  2. 4 puffs per day of long-acting rescue bronchodilator, or
  3. 2 nebulizer treatments per day.
* Subject has a post-bronchodilator FEV1 of less than 65% of predicted.
* Subject had three or more hospitalizations for exacerbations of asthma in the prior 12 months.
* Subject has a recent history of life-threatening asthma, defined by at least one intubation for asthma within the past five years.
* Subject had an ICU admission for asthma within the prior 24 months.
* Subject had four or more infections of the lower respiratory tract requiring antibiotics in the prior 12 months.
* Subject had four or more asthma exacerbations requiring oral steroid pulses in the prior 12 months.
* Subject has a known sensitivity to medications required to perform bronchoscopy (such as lidocaine, atropine, benzodiazepines, or other parasympathomimetic agents).
* Subject is undergoing immunosuppressant therapy other than steroids (e.g., methotrexate).
* Subject uses systemic beta-adrenergic blocking agents.
* Subject is an insulin-dependent diabetic.
* Subject is pregnant or a nursing mother, or has plans to become pregnant within the next 12 months.
* Subject has other respiratory diseases including interstitial lung disease, emphysema, cystic fibrosis, vocal cord dysfunction, mechanical upper airway obstruction, Churg-Strauss syndrome, or active allergic bronchopulmonary aspergillosis (current total IgE of >1000 Units/mL with positive specific IgE to aspergillus and evidence of central bronchiectasis).
* Subject has significant segmental atelectasis, lobar consolidation, significant or unstable pulmonary infiltrate, or pneumothorax, confirmed on X-ray.
* Subject has chronic sinus disease as defined by five or more episodes of sinusitis in past 12 months, or continuous symptoms of sinus infection (purulent discharge) and significant change in nasal steroid dosage in last six weeks.
* Subject has uncontrolled sleep apnea (sleep apnea not controlled by either dental appliances or continuous airway positive pressure (CPAP)).
* Subject has uncontrolled gastro-esophageal reflux disease as defined by a significant increase in therapy in last six weeks.
* Subject has lung cancer or a history of lung cancer.
* Subject currently has active cancer or a history of cancer with less than 5 years disease free survival time (whether or not there is evidence of local recurrence or metastases). Localized basal cell carcinoma (without metastases) of the skin is acceptable.

(Subject with a history of cancer (excluding lung cancer) and a five year or more disease free survival time may only be included in this Study by agreement of Sponsor on a case by case basis).

* Subject has a history of epilepsy.
* Subject currently has clinically significant cardiovascular or neurovascular disease, including myocardial infarction with congestive heart failure, angina, clinically significant cardiac dysrhythmia or conduction defect, cardiomegaly, cardiomyopathy, aortic aneurysm, cerebral vascular disease, or stroke.
* Subject is on anticoagulant therapy, has a bleeding diathesis, platelet dysfunction, or thrombocytopenia with platelet count less than 125,000/mm2 or known coagulopathy (INR > 1.5).
* Subject has uncontrolled hypertension (>200mm Hg systolic or >100mm Hg diastolic pressure).
* Subject has an electrical stimulation device such as a pacemaker, defibrillator, or deep nerve or deep brain stimulator.
* Subject has a psychiatric disorder that in the judgment of the Investigator could interfere with provision of Informed Consent, completion of tests, therapy, or follow-up visits.
* Subject has any other medical condition that in the Investigator's opinion would make them inappropriate for Study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Adverse Event Profile | 3 Months

IPD SHARING:
Plan to Share IPD: No
This study was cancelled prior to initiation.